CLINICAL TRIAL: NCT02197104
Title: Phase 2 Study of Citocoline for Treatment in Fragile X-associated Tremor/Ataxia Syndrome
Brief Title: Citocoline for Treatment in Fragile X-associated Tremor/Ataxia Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Deborah Hall, MD, Associate Professor Neurological Sciences, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CITO-123
Record Dates: First submitted 2014-07-14; First posted 2014-07-22 (Estimated); Results first posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Fragile X Tremor/Ataxia Syndrome
MeSH Terms: conditions — Fragile X Tremor Ataxia Syndrome | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Citocoline (Experimental): The intervention will be 1000mg of citicoline in capsule form once daily.
  Interventions: Drug: citocoline

INTERVENTIONS:
Drug: citocoline — Ten subjects will receive 1,000mg once daily of citicoline. Each subject will stay on the study drug for 12 months. The outcome measures will be assessed at baseline and then again at the end of month 3, month 6, and month 12. The subjects will continue taking the same study drug at the same dose throughout the entire trial.
  Other Names: CDP-choline

SUMMARY:
The objective of this study is to determine if citocoline is effective for balance abnormalities and to stabilize cognitive decline in patients with fragile X-associated tremor ataxia syndrome. The study will test 1000mg twice daily of citocoline for 12 months in an open label pilot study, with study visits at baseline, 3, 6, and 12 months.

DETAILED DESCRIPTION:
The purpose of this study was to determine if citicoline was safe for the treatment of tremor and balance abnormalities and to stabilize cognitive decline in patients with fragile X-associated tremor ataxia syndrome. Ten participants with diagnosed FXTAS were administered 1000 mg of citicoline once daily for 12 months. Outcome measures and neurological examination were performed at baseline, 3 months, 6 months, and 12 months. The primary outcome was safety. Secondary outcomes included change in FXTAS Rating Scale score, a battery of neuropsychological tests, an instrumented Timed up and go test, computerized dynamic posturography, 9-hole pegboard test, and balance confidence and psychiatric symptom questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of FXTAS

  * Serum creatine kinase, complete metabolic panel, complete blood count, liver function tests, renal function tests, platelets and EKG are within normal limits

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Presence of severe renal disease (BUN 50% greater than normal or creatinine clearance <60 mL/min) or hepatic disease.
* Abnormal creatine kinase and/or platelet count in the past 6 months (as determined by lab reports obtained from primary care physicians or conducted at baseline).
* Women of childbearing potential who are pregnant at the time of screening or who will not use adequate protection during participation of the study.
* Allergy/sensitivity to the drug of its formulations.
* Concurrent participation in another clinical study.
* Active substance use or dependence.
* Serious illness (requiring systematic treatment/or hospitalization) until the subject either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 60 days prior to study entry.
* Inability or unwillingness of the subject or legal guardian/representative to give written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Hall, MD PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Hall DA, Robertson EE, Leehey M, McAsey A, Ouyang B, Berry-Kravis E, O'Keefe JA. Open-label pilot clinical trial of citicoline for fragile X-associated tremor/ataxia syndrome (FXTAS). PLoS One. 2020 Feb 13;15(2):e0225191. doi: 10.1371/journal.pone.0225191. eCollection 2020. PMID 32053612

RESULTS

PARTICIPANT FLOW:
Groups:
- Citocoline: All participants received 1,000mg once daily of citicoline. Each subject will stay on the study drug for 12 months. The outcome measures will be assessed at baseline and then again at the end of month 3, month 6, and month 12. The subjects will continue taking the same study drug at the same dose throughout the entire trial.
Period: Overall Study
Arm/Group | Citocoline
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Citocoline: All participants were white and non-Hispanic; there were nine men and one woman. This distribution is expected as there is a lower penetrance of FXTAS in women from X-inactivation. The subject with probable FXTAS was also the female subject. Nine participants completed the one-year follow-up and one participant with a low platelet count withdrew prior to the end of the study and outcome data was missing for this participant at 12 months, but all available data were used for analysis.
Arm/Group | Citocoline
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (7.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Midwestern | 9
  United States: East Coast | 1

OUTCOME MEASURES:

1. Primary Outcome: FXTAS Rating Scale Score
Description: The FXTAS Rating Scale (FXTAS-RS), which was designed to measure the severity of motor signs in FXTAS patients, was administered to each participant. The FXTAS-RS was designed to measure the severity of motor signs of FXTAS, tremor, ataxia, and parkinsonism. The scale was developed from a combination of three separate measures: the Clinical Rating Scale for Tremor (CRST), the International Cooperative Ataxia Rating Scale (ICARS), and the Unified Parkinson's Disease Rating Scale (UPDRS). The resultant scale has 44 items and a possible total score of 0-226. A higher score indicates worse symptoms. For this study, improvement was defined as a 20% improvement on the FXTAS-RS.
Time Frame: 12 months
Population: 9 patients with FXTAS who participated in the study for 12 months were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Citocoline: Experimental group given the study drug, citocoline
Arm/Group | Citocoline
Number analyzed (Participants) | 9
score on a scale | 45.8 (21.22)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse event information was collected at baseline and then again at the end of month 3, month 6, and month 12.
Groups:
- Citocoline: All participants received citocoline.
Arm/Group | Citocoline
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 6/10
Other Adverse Events (participants affected / at risk) | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citocoline (N=10)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2) — Diarrhea, vomiting, elevated liver enzymes
Falls (Nervous system disorders) | 3 (3)
Low platelet count (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citocoline (N=10)
Bruising (Blood and lymphatic system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Leg edema (Blood and lymphatic system disorders) | 1 (1)
Weight gain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT02197104/Prot_SAP_000.pdf